CLINICAL TRIAL: NCT05308446
Title: Randomized Phase II Trial of Encorafenib and Cetuximab With or Without Nivolumab (NSC #748726) for Patients With Previously Treated, Microsatellite Stable, BRAFV600E Metastatic and/or Unresectable Colorectal Cancer
Brief Title: Testing the Addition of Nivolumab to Standard Treatment for Patients With Metastatic or Unresectable Colorectal Cancer That Have a BRAF Mutation
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2022-02494; NCI-2022-02494 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); S2107 (Other: SWOG); S2107 (Other: CTEP); U10CA180888 (NIH)
Record Dates: First submitted 2022-04-01; First posted 2022-04-04 (Actual); Last update posted 2025-09-18 (Actual); Status verified 2025-09

CONDITIONS: Metastatic Colon Adenocarcinoma; Metastatic Rectal Adenocarcinoma; Stage III Colon Cancer AJCC v8; Stage III Rectal Cancer AJCC v8; Stage IV Colon Cancer AJCC v8; Stage IV Rectal Cancer AJCC v8; Unresectable Colon Adenocarcinoma; Unresectable Rectal Adenocarcinoma
MeSH Terms: conditions — Colonic Neoplasms; Rectal Neoplasms | interventions — Cetuximab; (225)Ac-DOTA-c(RGDyK); encorafenib; Nivolumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm I (encorafenib, cetuximab, nivolumab) (Experimental): Patients receive encorafenib PO QD on days 1-28, cetuximab IV on days 1 and 15, and nivolumab IV on day 1. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: Cetuximab; Drug: Encorafenib; Biological: Nivolumab
- Arm II (encorafenib, cetuximab) (Active Comparator): Patients receive encorafenib PO QD on days 1-28 and cetuximab IV on days 1 and 15. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: Cetuximab; Drug: Encorafenib

INTERVENTIONS:
Biological: Cetuximab — Given IV
  Other Names: C 225; C-225; C225; Cetuximab Biosimilar CDP-1; Cetuximab Biosimilar CMAB009; Cetuximab Biosimilar KL 140; Chimeric Anti-EGFR Monoclonal Antibody; Chimeric MoAb C225; Chimeric Monoclonal Antibody C225; Erbitux; IMC-C225
Drug: Encorafenib — Given PO
  Other Names: Braftovi; LGX 818; LGX-818; LGX818
Biological: Nivolumab — Given IV
  Other Names: ABP 206; BCD-263; BMS 936558; BMS-936558; BMS936558; CMAB819; MDX 1106; MDX-1106; MDX1106; NIVO; Nivolumab Biosimilar ABP 206; Nivolumab Biosimilar BCD-263; Nivolumab Biosimilar CMAB819; ONO 4538; ONO-4538; ONO4538; Opdivo
  Arms: Arm I (encorafenib, cetuximab, nivolumab)

SUMMARY:
This phase II trial tests whether adding nivolumab to the usual treatment (encorafenib and cetuximab) works better than the usual treatment alone to shrink tumors in patients with colorectal cancer that has spread to other places in the body (metastatic) or that cannot be removed by surgery (unresectable) and whose tumor has a mutation in a gene called BRAF. Encorafenib is in a class of medications called kinase inhibitors. It is used in patients whose cancer has a certain mutation (change) in the BRAF gene. It works by blocking the action of mutated BRAF that signals cancer cells to multiply. This helps to stop or slow the spread of cancer cells. Cetuximab is in a class of medications called monoclonal antibodies. It binds to a protein called EGFR, which is found on some types of cancer cells. This may help keep cancer cells from growing. Immunotherapy with monoclonal antibodies, such as nivolumab, may help the body's immune system attack the cancer, and may interfere with the ability of tumor cells to grow and spread. Giving nivolumab in combination with encorafenib and cetuximab may be more effective than encorafenib and cetuximab alone at stopping tumor growth and spreading in patients with metastatic or unresectable BRAF-mutant colorectal cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To compare progression-free survival (PFS) per Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 in patients with microsatellite stable (MSS), BRAF^V600E metastatic and/or unresectable colorectal cancer (CRC) randomized to treatment with nivolumab + encorafenib + cetuximab compared to encorafenib + cetuximab.

SECONDARY OBJECTIVES:

I. To compare overall response rate (ORR), including confirmed and unconfirmed, complete and partial response, according to RECIST 1.1 criteria between the two arms.

II. To compare overall survival (OS) between the two arms. III. To compare duration of response between the two arms. IV. To compare safety and tolerability between the two arms. V. To assess immune-related PFS using modified response criteria adapted for immunotherapy (irRC-PFS) in patients treated with nivolumab + encorafenib + cetuximab.

BANKING OBJECTIVE:

I. To bank tissue and blood specimens for future correlative studies.

OUTLINE: Patients are randomized to 1 of 2 arms.

ARM I: Patients receive encorafenib orally (PO) once daily (QD) on days 1-28, cetuximab intravenously (IV) on days 1 and 15, and nivolumab IV on day 1. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.

ARM II: Patients receive encorafenib PO QD on days 1-28 and cetuximab IV on days 1 and 15. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed until death or 3 years after registration, whichever occurs first.

ELIGIBILITY:
Inclusion Criteria:

* Participants must have a histologically or cytologically confirmed diagnosis of adenocarcinoma of the colon or rectum. The date of diagnosis will be determined according to the pathologic date of diagnosis
* Participants must have measurable disease according to RECIST1.1 criteria. Computed tomography (CT) scans or magnetic resonance imaging (MRIs) used to assess measurable disease must have been completed within 28 days prior to registration. CT scans or MRIs used to assess non-measurable disease must have been completed within 42 days prior to registration. All disease must be assessed and documented on the Baseline Tumor Assessment Form
* Participants must have documented unresectable and/or metastatic disease on CT or MRI imaging. All disease must be assessed and documented on the Baseline Tumor Assessment Form
* Participants must have BRAF^V600E mutated colorectal cancer as tested in a Clinical Laboratory Improvement Act (CLIA)-certified laboratory
* Participants must have proficient mismatch repair (pMMR) or microsatellite stable (MSS) status as tested in a CLIA-certified laboratory and documented by the treating clinician. Proficient mismatch repair status can be determined by intact expression by immunohistochemistry of all 4 mismatch repair proteins (MLH1, MSH2, MSH6, and PMS2). Microsatellite instability can be determined by polymerase chain reaction (PCR)
* Participants with brain metastases must have completed surgery or radiation therapy >= 28 days prior to registration. These participants must have a CT or MRI of the brain showing no new or enlarging lesions within 42 days prior to registration. These participants must also be neurologically asymptomatic and without corticosteroid treatment for at least 7 days prior to registration. Metastatic brain parenchymal disease must have been treated and participant must be off steroids for 7 days prior to registration. The presence of leptomeningeal disease (LMD) is not considered stable disease, and participants with LMD are not eligible for this study
* Participants with known evidence of chronic hepatitis B virus (HBV) infection must have undetectable HBV viral load on suppressive therapy within 28 days prior to registration
* Participants with a history of hepatitis C virus (HCV) infection must have been treated and cured. Participants with HCV infection who are currently on treatment must have an undetectable HCV viral load within 28 days prior to registration
* Participants must have had one or two prior regimens of systemic chemotherapy for metastatic or locally advanced, unresectable disease. (A maintenance regimen of 5-fluorouracil or capecitabine, with or without bevacizumab, should not be counted as a separate line of treatment. The re-introduction of an initially successful induction regimen will not be counted as one additional line of treatment). Prior treatment for metastatic disease is not required for patients who experienced disease recurrence during or within 6 months of completion of adjuvant chemotherapy
* Participants must be of age >= 18 years at the time of informed consent
* Participants must have a Zubrod performance status of 0 or 1
* Participants must have a complete medical history and physical exam within 28 days prior to registration
* Absolute neutrophil count >= 1.0 x 10^3/uL (within 28 days prior to registration)
* Hemoglobin >= 9 g/dL (within 28 days prior to registration)
* Platelets >= 75 x 10^3/uL (within 28 days prior to registration)
* Total bilirubin =< 1.5 x institutional upper limit of normal (ULN) (within 28 days prior to registration)
* Aspartate aminotransferase (AST)/alanine aminotransferase (ALT) =< 3 x institutional ULN (within 28 days prior to registration)
* If liver metastases are present, then it is acceptable for AST level =< 5.0 x ULN, and/or an ALT level =< 5.0 x ULN (within 28 days prior to registration)
* Participants must have serum creatinine =< the IULN OR measured OR calculated creatinine clearance >= 50 mL/min using the Cockroft-Gault Formula. This specimen must have been drawn and processed within 28 days prior to registration
* Participants must be able to swallow and retain pills
* Participants must have adequate cardiac function. Participants with known history or current symptoms of cardiac disease, or history of treatment with cardiotoxic agents, must have a clinical risk assessment of cardiac function using the New York Heart Association Functional Classification. To be eligible for this trial, participants must be class 2 or better
* Participants with a known significant risk of corrected QT interval (QTc) prolongation must have an electrocardiogram (ECG) performed within 28 days prior to prior to registration

  * Note: Per package insert for encorafenib, participants already at risk for development of QTc prolongation include those who "already have or who are at significant risk of developing QTc prolongation, including participants with known long QT syndromes, clinically significant bradyarrhythmias, severe or uncontrolled heart failure and those taking other medicinal products associated with QT prolongation."
* Participants must be offered the opportunity to participate in specimen banking. With participant consent, specimens must be collected and submitted via the Southwest Oncology Group (SWOG) Specimen Tracking System
* Participants must be informed of the investigational nature of this study and must sign and give informed consent in accordance with institutional and federal guidelines.

  * Note: As a part of the OPEN registration process, the treating institution's identity is provided in order to ensure that the current (within 365 days) date of institutional review board approval for this study has been entered in the system

Exclusion Criteria:

* Participants must not have a known positive serology for human immunodeficiency virus (HIV). Encorafenib is contraindicated with concomitant use of non-nucleoside analog reverse transcriptase inhibitors like efavirenz and etravirine. In addition, it is recommended in the investigator brochure of encorafenib to avoid using encorafenib with protease inhibitors. Therefore, because all participants on this study would receive encorafenib for either randomized arm of treatment, participants with HIV who receive these components of highly active antiretroviral therapy (HAART) would be at high risk for complications of drug-drug interaction
* Participants must not have had prior treatment with a BRAF inhibitor (including, but not limited to, encorafenib, dabrafenib, or vemurafenib), MEK inhibitor (including, but not limited to, trametinib, selumetinib, or binimetinib), or ERK inhibitor (of note, regorafenib is not considered a BRAF inhibitor for the context of eligibility criteria)
* Participants must not have had prior treatment with anti-EGFR therapies
* Participants must not have had prior treatment with an anti-PD-1, anti-PD-L1, anti-PD-L2, anti-CTLA-4 antibody, or any other antibody or drug specifically targeting T-cell co-stimulation or immune checkpoint pathways
* Participants must not have a condition requiring systemic treatment with either corticosteroids (> 10 mg daily prednisone equivalents) or other immunosuppressive medications within 14 days of registration. Inhaled or topical steroids and adrenal replacement doses < 10 mg daily prednisone equivalents are permitted in the absence of active autoimmune disease. Patients are permitted to use topical, ocular, intra-articular, intranasal, and inhalational corticosteroids (with minimal systemic absorption). Physiologic replacement doses of systemic corticosteroids are permitted, even if < 10 mg/day prednisone equivalents. A brief course of corticosteroids for prophylaxis (e.g., contrast dye allergy) or for treatment of non-autoimmune conditions (e.g., delayed-type hypersensitivity reaction caused by contact allergen) is permitted, as long as there has been a washout period for corticosteroids of >= 7 days prior to registration
* Participants must not have received a live vaccine within 30 days prior to study registration. Seasonal flu and COVID vaccines that do not contain a live virus are permitted
* Participants must not be receiving any other investigational agents
* Participants must not have impaired gastrointestinal function or disease that may significantly alter the absorption of study drug (e.g., ulcerative diseases, uncontrolled vomiting, malabsorption syndrome, small bowel resection with decreased intestinal absorption)
* Participants must not have a history of inflammatory bowel disease, (including ulcerative colitis and Crohn's disease), symptomatic autoimmune disease (e.g., rheumatoid arthritis, systemic progressive sclerosis [scleroderma], systemic lupus erythematosus, autoimmune vasculitis [e.g., Wegener's Granulomatosis]); central nervous system (CNS) or motor neuropathy considered of autoimmune origin (e.g., Guillain-Barre Syndrome and myasthenia gravis, multiple sclerosis).

  * Note: Participants with Graves' disease will be allowed
* Participants must not have a history of pneumonitis that has required oral or intravenous (IV) steroids within the last 12 months
* Participants must not have a history of a grade 3 or 4 allergic reaction attributed to humanized or human monoclonal antibody therapy
* Participants must not have a history of a prior allogeneic tissue or solid organ transplant
* Participants must not have a history of acute coronary syndromes (including myocardial infarction, unstable angina, coronary artery bypass grafting, coronary angioplasty, or stenting) within 6 months prior to study registration
* Participants must not have uncontrolled blood pressure and hypertension within 28 days prior to registration.

  * Uncontrolled blood pressure and hypertension is defined as systolic blood pressure (SBP) >= 160 mmHg or diastolic blood pressure (DBP) > 100 mmHg within 28 days prior to registration. Participants are permitted to be receiving multiple anti-hypertensive medications (unless otherwise indicated in the study). All blood pressure measurements within the 28 days prior to registration must be SBP < 160 and DBP =< 100. An exception can be made by a healthcare provider for a participant with a single blood pressure elevation who upon rechecking has a normal blood pressure
* Participants must not have a prior or concurrent malignancy whose natural history or treatment (in the opinion of the treating physician) has the potential to interfere with the safety or efficacy assessment of the investigational regimen or requires concurrent therapy
* Participants must not be pregnant or nursing. Individuals who are of reproductive potential must have agreed to use an effective contraceptive method with details provided as a part of the consent process. A person who has had menses at any time in the preceding 12 consecutive months or who has semen likely to contain sperm is considered to be of "reproductive potential." In addition to routine contraceptive methods, "effective contraception" also includes refraining from sexual activity that might result in pregnancy and surgery intended to prevent pregnancy (or with a side-effect of pregnancy prevention) including hysterectomy, bilateral oophorectomy, bilateral tubal ligation/occlusion and vasectomy with testing showing no sperm in the semen
* Participants must not be planning treatment with other systemic anti-cancer agents (e.g., chemotherapy, hormonal therapy, immunotherapy) or other treatments not part of protocol-specified anti-cancer therapy including concurrent investigational agents of any type

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Estimated)
Dates: Start 2022-07-19 (Actual); Primary Completion 2026-02-28 (Estimated); Study Completion 2026-02-28 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival (PFS) | From date of registration to date of first documentation of progression or symptomatic deterioration, or death due to any cause, assessed up to 3 years
  Conducted in all eligible participants according to the intent-to-treat principle using the stratified log rank test when a total of 66 PFS events have been observed. Estimated using the Kaplan-Meier method and compared using the stratified log rank test.

SECONDARY OUTCOMES:
Overall response rate (ORR) | Up to 3 years
  Evaluated per Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 (confirmed and unconfirmed, complete and partial response) and compared across treatment arms via Fisher's exact test.
Overall survival (OS) | From date of registration to date of death due to any cause, assessed up to 3 years
  Estimated using the Kaplan-Meier method and compared using the stratified log rank test. The distribution of OS will be estimated using the method of Kaplan-Meier and compared using the stratified log rank test.
Duration of response (DoR) | From date of first documentation of confirmed response (complete response or partial response) to date of first documentation of progression or symptomatic deterioration or death due to any cause among participants who achieve a response, up to 3 years
  Estimated using the Kaplan-Meier method and compared using the stratified log rank test. The distribution of DoR will be estimated using the method of Kaplan-Meier and compared using the stratified log rank test.
Immune related progression-free survival (irRC-PFS) in Arm I | From date of registration to date of initial documentation of irRC-progression that has subsequently been confirmed or symptomatic deterioration, or death due to any cause, assessed up to 3 years
  The distribution of irRC-PFS in Arm 1 (nivolumab + encorafenib + cetuximab) will be estimated using the method of Kaplan-Meier.
Incidence of adverse events | Up to 3 years
  At least 25 eligible participants in each arm are sufficient to estimate the probability of a particular toxicity within ±20% (95% confidence interval), and any toxicity occurring with at least 10% probability is likely (93% chance) to be seen at least once. At least 50 eligible participants are sufficient to estimate the probability of a particular toxicity within ±14% (95% confidence interval), and any toxicity occurring with at least 5% probability is likely (92% chance) to be seen at least once.

CONTACTS AND LOCATIONS:
Overall Officials: Van K Morris, Principal Investigator — SWOG Cancer Research Network
Locations (286):
- United States (282):
  - CTCA at Western Regional Medical Center, Goodyear, Arizona
  - Mercy Cancer Center - Carmichael, Carmichael, California
  - Mercy San Juan Medical Center, Carmichael, California
  - Kaiser Permanente Dublin, Dublin, California
  - Mercy Cancer Center - Elk Grove, Elk Grove, California
  - Kaiser Permanente-Fremont, Fremont, California
  - Kaiser Permanente-Fresno, Fresno, California
  - UCI Health - Chao Family Comprehensive Cancer Center and Ambulatory Care, Irvine, California
  - Kaiser Permanente-Modesto, Modesto, California
  - Kaiser Permanente-Oakland, Oakland, California
  - UC Irvine Health/Chao Family Comprehensive Cancer Center, Orange, California
  - Mercy Cancer Center - Rocklin, Rocklin, California
  - Kaiser Permanente-Roseville, Roseville, California
  - Kaiser Permanente Downtown Commons, Sacramento, California
  - Mercy Cancer Center - Sacramento, Sacramento, California
  - Kaiser Permanente-South Sacramento, Sacramento, California
  - Kaiser Permanente-San Francisco, San Francisco, California
  - Kaiser Permanente-Santa Teresa-San Jose, San Jose, California
  - Kaiser Permanente San Leandro, San Leandro, California
  - Kaiser Permanente Medical Center - Santa Clara, Santa Clara, California
  - Kaiser Permanente-Santa Rosa, Santa Rosa, California
  - Kaiser Permanente-South San Francisco, South San Francisco, California
  - Kaiser Permanente-Vallejo, Vallejo, California
  - Kaiser Permanente-Walnut Creek, Walnut Creek, California
  - Woodland Memorial Hospital, Woodland, California
  - UCHealth University of Colorado Hospital, Aurora, Colorado
  - Rocky Mountain Cancer Centers-Penrose, Colorado Springs, Colorado
  - UCHealth Memorial Hospital Central, Colorado Springs, Colorado
  - Memorial Hospital North, Colorado Springs, Colorado
  - Poudre Valley Hospital, Fort Collins, Colorado
  - Cancer Care and Hematology-Fort Collins, Fort Collins, Colorado
  - UCHealth Greeley Hospital, Greeley, Colorado
  - UCHealth Highlands Ranch Hospital, Highlands Ranch, Colorado
  - Medical Center of the Rockies, Loveland, Colorado
  - CTCA at Southeastern Regional Medical Center, Newnan, Georgia
  - Kaiser Permanente Moanalua Medical Center, Honolulu, Hawaii
  - Saint Alphonsus Cancer Care Center-Boise, Boise, Idaho
  - Saint Luke's Cancer Institute - Boise, Boise, Idaho
  - Saint Alphonsus Cancer Care Center-Caldwell, Caldwell, Idaho
  - Kootenai Health - Coeur d'Alene, Coeur d'Alene, Idaho
  - Saint Luke's Cancer Institute - Fruitland, Fruitland, Idaho
  - Saint Luke's Cancer Institute - Meridian, Meridian, Idaho
  - Saint Alphonsus Cancer Care Center-Nampa, Nampa, Idaho
  - Saint Luke's Cancer Institute - Nampa, Nampa, Idaho
  - Kootenai Clinic Cancer Services - Post Falls, Post Falls, Idaho
  - Kootenai Clinic Cancer Services - Sandpoint, Sandpoint, Idaho
  - Saint Luke's Cancer Institute - Twin Falls, Twin Falls, Idaho
  - Rush-Copley Medical Center, Aurora, Illinois
  - Advocate Good Shepherd Hospital, Barrington, Illinois
  - Illinois CancerCare-Bloomington, Bloomington, Illinois
  - Illinois CancerCare-Canton, Canton, Illinois
  - Illinois CancerCare-Carthage, Carthage, Illinois
  - Centralia Oncology Clinic, Centralia, Illinois
  - University of Illinois, Chicago, Illinois
  - Advocate Illinois Masonic Medical Center, Chicago, Illinois
  - AMG Crystal Lake - Oncology, Crystal Lake, Illinois
  - Carle at The Riverfront, Danville, Illinois
  - Cancer Care Specialists of Illinois - Decatur, Decatur, Illinois
  - Decatur Memorial Hospital, Decatur, Illinois
  - Illinois CancerCare-Dixon, Dixon, Illinois
  - Advocate Good Samaritan Hospital, Downers Grove, Illinois
  - Carle Physician Group-Effingham, Effingham, Illinois
  - Crossroads Cancer Center, Effingham, Illinois
  - Advocate Sherman Hospital, Elgin, Illinois
  - Illinois CancerCare-Eureka, Eureka, Illinois
  - Illinois CancerCare-Galesburg, Galesburg, Illinois
  - Advocate South Suburban Hospital, Hazel Crest, Illinois
  - Illinois CancerCare-Kewanee Clinic, Kewanee, Illinois
  - AMG Libertyville - Oncology, Libertyville, Illinois
  - Condell Memorial Hospital, Libertyville, Illinois
  - Illinois CancerCare-Macomb, Macomb, Illinois
  - Carle Physician Group-Mattoon/Charleston, Mattoon, Illinois
  - Cancer Care Center of O'Fallon, O'Fallon, Illinois
  - Advocate Christ Medical Center, Oak Lawn, Illinois
  - Illinois CancerCare-Ottawa Clinic, Ottawa, Illinois
  - Advocate Lutheran General Hospital, Park Ridge, Illinois
  - Illinois CancerCare-Pekin, Pekin, Illinois
  - Illinois CancerCare-Peoria, Peoria, Illinois
  - Illinois CancerCare-Peru, Peru, Illinois
  - Illinois CancerCare-Princeton, Princeton, Illinois
  - Southern Illinois University School of Medicine, Springfield, Illinois
  - Springfield Clinic, Springfield, Illinois
  - Springfield Memorial Hospital, Springfield, Illinois
  - Carle Cancer Center, Urbana, Illinois
  - Illinois CancerCare - Washington, Washington, Illinois
  - Rush-Copley Healthcare Center, Yorkville, Illinois
  - Northwest Cancer Center - Main Campus, Crown Point, Indiana
  - Northwest Oncology LLC, Dyer, Indiana
  - Northwest Cancer Center - Hobart, Hobart, Indiana
  - Saint Mary Medical Center, Hobart, Indiana
  - Franciscan Health Indianapolis, Indianapolis, Indiana
  - Saint Catherine Hospital, Indianapolis, Indiana
  - Franciscan Saint Elizabeth Health - Lafayette East, Lafayette, Indiana
  - Woodland Cancer Care Center, Michigan City, Indiana
  - Franciscan Health Mooresville, Mooresville, Indiana
  - The Community Hospital, Munster, Indiana
  - Women's Diagnostic Center - Munster, Munster, Indiana
  - Northwest Cancer Center - Valparaiso, Valparaiso, Indiana
  - Mary Greeley Medical Center, Ames, Iowa
  - McFarland Clinic - Ames, Ames, Iowa
  - McFarland Clinic - Boone, Boone, Iowa
  - Mercy Medical Center - Des Moines, Des Moines, Iowa
  - McFarland Clinic - Trinity Cancer Center, Fort Dodge, Iowa
  - McFarland Clinic - Jefferson, Jefferson, Iowa
  - McFarland Clinic - Marshalltown, Marshalltown, Iowa
  - LSU Health Baton Rouge-North Clinic, Baton Rouge, Louisiana
  - Our Lady of the Lake Physician Group, Baton Rouge, Louisiana
  - Ochsner Hematology Oncology North Shore - Covington (West Region), Covington, Louisiana
  - Ochsner Medical Center Jefferson, New Orleans, Louisiana
  - Trinity Health Saint Joseph Mercy Hospital Ann Arbor, Ann Arbor, Michigan
  - Bronson Battle Creek, Battle Creek, Michigan
  - Trinity Health IHA Medical Group Hematology Oncology - Brighton, Brighton, Michigan
  - Trinity Health Medical Center - Brighton, Brighton, Michigan
  - Trinity Health IHA Medical Group Hematology Oncology - Canton, Canton, Michigan
  - Trinity Health Medical Center - Canton, Canton, Michigan
  - Chelsea Hospital, Chelsea, Michigan
  - Trinity Health IHA Medical Group Hematology Oncology - Chelsea Hospital, Chelsea, Michigan
  - Henry Ford Hospital, Detroit, Michigan
  - Henry Ford Health Saint John Hospital, Detroit, Michigan
  - Henry Ford River District Hospital, East China Township, Michigan
  - Cancer Hematology Centers - Flint, Flint, Michigan
  - Genesee Hematology Oncology PC, Flint, Michigan
  - Genesys Hurley Cancer Institute, Flint, Michigan
  - Hurley Medical Center, Flint, Michigan
  - Corewell Health Grand Rapids Hospitals - Butterworth Hospital, Grand Rapids, Michigan
  - Trinity Health Grand Rapids Hospital, Grand Rapids, Michigan
  - Henry Ford Saint John Hospital - Academic, Grosse Pointe Woods, Michigan
  - Henry Ford Saint John Hospital - Van Elslander, Grosse Pointe Woods, Michigan
  - Bronson Methodist Hospital, Kalamazoo, Michigan
  - West Michigan Cancer Center, Kalamazoo, Michigan
  - Beacon Kalamazoo Cancer Center, Kalamazoo, Michigan
  - University of Michigan Health - Sparrow Lansing, Lansing, Michigan
  - Trinity Health Saint Mary Mercy Livonia Hospital, Livonia, Michigan
  - Henry Ford Saint John Hospital - Macomb Medical, Macomb, Michigan
  - Trinity Health Muskegon Hospital, Muskegon, Michigan
  - Corewell Health Lakeland Hospitals - Niles Hospital, Niles, Michigan
  - Cancer and Hematology Centers of Western Michigan - Norton Shores, Norton Shores, Michigan
  - Henry Ford Health Providence Novi Hospital, Novi, Michigan
  - Henry Ford Medical Center-Columbus, Novi, Michigan
  - Corewell Health Reed City Hospital, Reed City, Michigan
  - MyMichigan Medical Center Saginaw, Saginaw, Michigan
  - Oncology Hematology Associates of Saginaw Valley PC, Saginaw, Michigan
  - Corewell Health Lakeland Hospitals - Marie Yeager Cancer Center, Saint Joseph, Michigan
  - Henry Ford Health Providence Southfield Hospital, Southfield, Michigan
  - Bhadresh Nayak MD PC-Sterling Heights, Sterling Heights, Michigan
  - MyMichigan Medical Center Tawas, Tawas City, Michigan
  - Munson Medical Center, Traverse City, Michigan
  - Henry Ford Health Warren Hospital, Warren, Michigan
  - Henry Ford Warren Hospital - GLCMS, Warren, Michigan
  - Macomb Hematology Oncology PC, Warren, Michigan
  - Henry Ford West Bloomfield Hospital, West Bloomfield, Michigan
  - Saint Mary's Oncology/Hematology Associates of West Branch, West Branch, Michigan
  - University of Michigan Health - West, Wyoming, Michigan
  - Huron Gastroenterology PC, Ypsilanti, Michigan
  - Trinity Health IHA Medical Group Hematology Oncology Ann Arbor Campus, Ypsilanti, Michigan
  - Mercy Hospital, Coon Rapids, Minnesota
  - Essentia Health - Deer River Clinic, Deer River, Minnesota
  - Essentia Health Cancer Center, Duluth, Minnesota
  - Fairview Southdale Hospital, Edina, Minnesota
  - Essentia Health Hibbing Clinic, Hibbing, Minnesota
  - Abbott-Northwestern Hospital, Minneapolis, Minnesota
  - North Memorial Medical Health Center, Robbinsdale, Minnesota
  - Park Nicollet Clinic - Saint Louis Park, Saint Louis Park, Minnesota
  - Regions Hospital, Saint Paul, Minnesota
  - United Hospital, Saint Paul, Minnesota
  - Essentia Health Sandstone, Sandstone, Minnesota
  - Essentia Health Virginia Clinic, Virginia, Minnesota
  - Saint Francis Medical Center, Cape Girardeau, Missouri
  - Community Hospital of Anaconda, Anaconda, Montana
  - Billings Clinic Cancer Center, Billings, Montana
  - Bozeman Health Deaconess Hospital, Bozeman, Montana
  - Benefis Sletten Cancer Institute, Great Falls, Montana
  - Logan Health Medical Center, Kalispell, Montana
  - Community Medical Center, Missoula, Montana
  - Dartmouth Hitchcock Medical Center/Dartmouth Cancer Center, Lebanon, New Hampshire
  - Hunterdon Medical Center, Flemington, New Jersey
  - Roswell Park Cancer Institute, Buffalo, New York
  - Southeastern Medical Oncology Center-Clinton, Clinton, North Carolina
  - Southeastern Medical Oncology Center-Goldsboro, Goldsboro, North Carolina
  - Southeastern Medical Oncology Center-Jacksonville, Jacksonville, North Carolina
  - FirstHealth of the Carolinas-Moore Regional Hospital, Pinehurst, North Carolina
  - Strecker Cancer Center-Belpre, Belpre, Ohio
  - Miami Valley Hospital South, Centerville, Ohio
  - Adena Regional Medical Center, Chillicothe, Ohio
  - Mount Carmel East Hospital, Columbus, Ohio
  - Columbus Oncology and Hematology Associates Inc, Columbus, Ohio
  - Riverside Methodist Hospital, Columbus, Ohio
  - Grant Medical Center, Columbus, Ohio
  - The Mark H Zangmeister Center, Columbus, Ohio
  - Doctors Hospital, Columbus, Ohio
  - Miami Valley Hospital, Dayton, Ohio
  - Premier Blood and Cancer Center, Dayton, Ohio
  - Dayton Physician LLC - Englewood, Dayton, Ohio
  - Miami Valley Hospital North, Dayton, Ohio
  - Delaware Health Center-Grady Cancer Center, Delaware, Ohio
  - Grady Memorial Hospital, Delaware, Ohio
  - Columbus Oncology and Hematology Associates, Dublin, Ohio
  - Atrium Medical Center-Middletown Regional Hospital, Franklin, Ohio
  - Dayton Physicians LLC-Atrium, Franklin, Ohio
  - Miami Valley Cancer Care and Infusion, Greenville, Ohio
  - Mount Carmel Grove City Hospital, Grove City, Ohio
  - Kettering Medical Center, Kettering, Ohio
  - Fairfield Medical Center, Lancaster, Ohio
  - OhioHealth Mansfield Hospital, Mansfield, Ohio
  - OhioHealth Marion General Hospital, Marion, Ohio
  - Memorial Hospital, Marysville, Ohio
  - Knox Community Hospital, Mount Vernon, Ohio
  - Licking Memorial Hospital, Newark, Ohio
  - Southern Ohio Medical Center, Portsmouth, Ohio
  - Springfield Regional Cancer Center, Springfield, Ohio
  - Springfield Regional Medical Center, Springfield, Ohio
  - Toledo Clinic Cancer Centers-Toledo, Toledo, Ohio
  - Upper Valley Medical Center, Troy, Ohio
  - Saint Ann's Hospital, Westerville, Ohio
  - Genesis Healthcare System Cancer Care Center, Zanesville, Ohio
  - Cancer Centers of Southwest Oklahoma Research, Lawton, Oklahoma
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Mercy Hospital Oklahoma City, Oklahoma City, Oklahoma
  - Clackamas Radiation Oncology Center, Clackamas, Oregon
  - Providence Cancer Institute Clackamas Clinic, Clackamas, Oregon
  - Providence Newberg Medical Center, Newberg, Oregon
  - Saint Alphonsus Cancer Care Center-Ontario, Ontario, Oregon
  - Providence Willamette Falls Medical Center, Oregon City, Oregon
  - Providence Portland Medical Center, Portland, Oregon
  - Providence Saint Vincent Medical Center, Portland, Oregon
  - Lehigh Valley Hospital-Cedar Crest, Allentown, Pennsylvania
  - Lehigh Valley Hospital - Muhlenberg, Bethlehem, Pennsylvania
  - University of Pennsylvania/Abramson Cancer Center, Philadelphia, Pennsylvania
  - Reading Hospital, West Reading, Pennsylvania
  - Rhode Island Hospital, Providence, Rhode Island
  - Prisma Health Cancer Institute - Spartanburg, Boiling Springs, South Carolina
  - Medical University of South Carolina, Charleston, South Carolina
  - Prisma Health Cancer Institute - Easley, Easley, South Carolina
  - Prisma Health Cancer Institute - Butternut, Greenville, South Carolina
  - Prisma Health Cancer Institute - Faris, Greenville, South Carolina
  - Prisma Health Greenville Memorial Hospital, Greenville, South Carolina
  - Prisma Health Cancer Institute - Eastside, Greenville, South Carolina
  - Prisma Health Cancer Institute - Greer, Greer, South Carolina
  - Prisma Health Cancer Institute - Seneca, Seneca, South Carolina
  - Vanderbilt University/Ingram Cancer Center, Nashville, Tennessee
  - The Don and Sybil Harrington Cancer Center, Amarillo, Texas
  - UT Southwestern Simmons Cancer Center - RedBird, Dallas, Texas
  - UT Southwestern/Simmons Cancer Center-Dallas, Dallas, Texas
  - UT Southwestern/Simmons Cancer Center-Fort Worth, Fort Worth, Texas
  - M D Anderson Cancer Center, Houston, Texas
  - UT Southwestern Clinical Center at Richardson/Plano, Richardson, Texas
  - Huntsman Cancer Institute/University of Utah, Salt Lake City, Utah
  - Dartmouth Cancer Center - North, Saint Johnsbury, Vermont
  - Swedish Cancer Institute-Edmonds, Edmonds, Washington
  - Swedish Cancer Institute-Issaquah, Issaquah, Washington
  - Swedish Medical Center-First Hill, Seattle, Washington
  - United Hospital Center, Bridgeport, West Virginia
  - West Virginia University Healthcare, Morgantown, West Virginia
  - ThedaCare Regional Cancer Center, Appleton, Wisconsin
  - Duluth Clinic Ashland, Ashland, Wisconsin
  - Aurora Cancer Care-Southern Lakes VLCC, Burlington, Wisconsin
  - Aurora Saint Luke's South Shore, Cudahy, Wisconsin
  - Marshfield Medical Center-EC Cancer Center, Eau Claire, Wisconsin
  - Aurora Health Care Germantown Health Center, Germantown, Wisconsin
  - Aurora Cancer Care-Grafton, Grafton, Wisconsin
  - Aurora BayCare Medical Center, Green Bay, Wisconsin
  - Aurora Cancer Care-Kenosha South, Kenosha, Wisconsin
  - Aurora Bay Area Medical Group-Marinette, Marinette, Wisconsin
  - Marshfield Medical Center-Marshfield, Marshfield, Wisconsin
  - Aurora Cancer Care-Milwaukee, Milwaukee, Wisconsin
  - Aurora Saint Luke's Medical Center, Milwaukee, Wisconsin
  - Aurora Sinai Medical Center, Milwaukee, Wisconsin
  - Marshfield Medical Center - Minocqua, Minocqua, Wisconsin
  - ProHealth D N Greenwald Center, Mukwonago, Wisconsin
  - Cancer Center of Western Wisconsin, New Richmond, Wisconsin
  - ProHealth Oconomowoc Memorial Hospital, Oconomowoc, Wisconsin
  - Vince Lombardi Cancer Clinic - Oshkosh, Oshkosh, Wisconsin
  - Aurora Cancer Care-Racine, Racine, Wisconsin
  - Marshfield Medical Center-Rice Lake, Rice Lake, Wisconsin
  - Vince Lombardi Cancer Clinic-Sheboygan, Sheboygan, Wisconsin
  - Marshfield Medical Center-River Region at Stevens Point, Stevens Point, Wisconsin
  - Aurora Medical Center in Summit, Summit, Wisconsin
  - Vince Lombardi Cancer Clinic-Two Rivers, Two Rivers, Wisconsin
  - UW Cancer Center at ProHealth Care, Waukesha, Wisconsin
  - Aurora Cancer Care-Milwaukee West, Wauwatosa, Wisconsin
  - Aurora West Allis Medical Center, West Allis, Wisconsin
  - Marshfield Medical Center - Weston, Weston, Wisconsin
- Puerto Rico (4):
  - Puerto Rico Hematology Oncology Group, Bayamón
  - Centro Comprensivo de Cancer de UPR, San Juan
  - PROncology, San Juan
  - San Juan City Hospital, San Juan

IPD SHARING:
Plan to Share IPD: Yes
"NCI is committed to sharing data in accordance with NIH policy. For more details on how clinical trial data is shared, access the link to the NIH data sharing policy page."
URL: https://grants.nih.gov/policy/sharing.htm

DOCUMENTS (1):
  • Informed Consent Form (2023-08-10): https://cdn.clinicaltrials.gov/large-docs/46/NCT05308446/ICF_000.pdf